CLINICAL TRIAL: NCT00361868
Title: A Randomized, Double-Blind Trial Comparing the Efficacy and Safety of a Fixed Combination of Fenofibrate and Metformin vs Rosiglitazone in Patients With Type 2 Diabetes Mellitus and Dyslipidemia
Brief Title: Fenofibrate and Metformin Fixed Combination vs Rosiglitazone - FAME ROSI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was discontinued prematurely at the end of March 2007 due to slow enrolment.
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Michel Conte, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C LF23-0121 05 01; 2005-006060-63
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Dyslipidemia; Glucose Metabolism Disorder
Keywords: Treatment of Dyslipidemia and of Type 2 Diabetes Mellitus
MeSH Terms: conditions — Dyslipidemias; Glucose Metabolism Disorders | interventions — Fenofibrate; Metformin; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: fenofibrate (F) + metformin (M) hydrochloride fixed combination
- 2 (Active Comparator)
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: fenofibrate (F) + metformin (M) hydrochloride fixed combination — First period: F80mg/M500mg - per os - twice a day during 2 weeks and F80mg/M850mg - per os - twice a day during 10 weeks - Second period: F54mg/M850mg - per os - three times a day during 12 weeks
  Arms: 1
Drug: Rosiglitazone — First period: 4 mg - per os - daily during 12 weeks - Second period: 4 mg - per os - twice a day during 12 weeks
  Arms: 2

SUMMARY:
Under conditions of first-line drug treatment in antidiabetic drug naïve/drug free patients with type 2 diabetes mellitus and dyslipidemia, to show that :- the efficacy of a fixed combination (FC) of fenofibrate and metformin on glycemic control is not inferior to that of rosiglitazone and the efficacy of FC of fenofibrate and metformin on triglyceride control is superior to that of rosiglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Type 2 diabetes mellitus and dyslipidemia inadequately controlled with lifestyle modifications.

Exclusion Criteria:

* Type 1 diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
HbA1c/TG | 24 weeks

SECONDARY OUTCOMES:
Lipid and glycemic parameters. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (70):
- Croatia (6):
  - Site105, Pula
  - Site102, Rijeka
  - Site103, Split
  - Site104, Varaždin
  - Site100, Zagreb
  - Site101, Zagreb
- Finland (4):
  - Site 205, Jyväskylä
  - Site 206, Kokkola
  - Site 208, Laukaa
  - Site 207, Oulu
- France (7):
  - Site 303, Bassens
  - Site 307, Bordeaux
  - Site 305, Mûrs-Erigné
  - Site 302, Seysses
  - Site 304, Strasbourg
  - Site 301, Thouars
  - Site 306, Vihiers
- Germany (14):
  - Site 405, Berlin
  - Site 410, Borna
  - Site 403, Bretten
  - Site 402, Dresden
  - Site 404, Frankfurt
  - Site 400, Freiburg im Breisgau
  - Site 401, Hanover
  - Site 409, Ilvesheim
  - Site 411, Ilvesheim
  - Site 407, Leipzig
  - Site 406, Rodgau
  - Site 413, Rotenburg (Wümme)
  - Site 408, Schwerin
  - Site 412, Villingen-Schwenningen
- Netherlands (9):
  - Site 509, Almere Stad
  - Site 502, Breda
  - Site 503, Eindhoven
  - Site 504, Groningen
  - Site 505, Leiden
  - Site 506, Nijmegen
  - Site 500, Rotterdam
  - Site 507, Velp
  - Site 508, Zoetermeer
- Poland (12):
  - Site 610, Bialystok
  - Site 606, Elblag
  - Site 608, Gdansk
  - Site 600, Lodz
  - Site 605, Otolinska
  - Site 604, Radom
  - Site 613, Starogard Gdański
  - Site 601, Warsaw
  - Site 607, Warsaw
  - Site 612, Warsaw
  - Site 602, Wroclaw
  - Site 603, Wroclaw
- Romania (6):
  - Site 704, Brasov
  - Site 701, Bucharest
  - Site 703, Bucharest
  - Site 700, Cluj-Napoca
  - Site 702, Iași
  - Site 705, Târgu Mureş
- Ukraine (12):
  - Site 807, Kharkiv
  - Site 811, Kharkiv
  - Site 812, Kharkiv
  - Site 800, Kiev
  - Site 803, Kiev
  - Site 808, Kiev
  - Site 809, Kiev
  - Site 810, Kiev
  - Site 813, Kiev
  - Site 805, Lviv
  - Site 804, Odesa
  - Site 802, Vinnitsa